CLINICAL TRIAL: NCT00255060
Title: Comprehensive Screening for Women at High Genetic Risk for Developing Breast Cancer
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); United States Department of Defense (U.S. Federal Agency)
Responsible Party: James M Ford, Stanford University School of Medicine
Other Study IDs: BRSNSTU0002; 77716; BRSNSTU0002; NCT00255060
Record Dates: First submitted 2005-11-15; First posted 2005-11-17 (Estimated); Last update posted 2010-07-20 (Estimated); Status verified 2010-07

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
To screen women who are high risk for breast cancer with breast MRI, mammogram and random periareolar fine needle aspiration.

DETAILED DESCRIPTION:
General Purpose: The purpose of our protocol is develop a comprehensive screening protocol for women at high risk for developing breast cancer in the hopes of detecting breast cancer or it's precursor lesions at the earliest possible stage and reducing breast cancer mortality.

The following are our specific goals in this endeavor;

1. To assess the sensitivity and specificity of MRI in breast cancer detection in women at high risk compared to mammography
2. To assess the ability of random periareolar fine needle aspiration to detect abnormal ductal cells and to correlate these results with MRI and mammogram findings
3. To assess appropriate screening intervals for BRCA1/2 mutation carriers and women with a >10% risk of developing breast cancer in ten years The following aims will be outlined in detail under methodology.

ELIGIBILITY:
Inclusion Criteria:Subjects must be female, between the ages of 25 and 65, or ten years younger than the youngest breast cancer diagnosed in the family, or have no mutation identified but have a greater than 10% risk of developing breast cancer in ten years (based on the Claus Model).

May have had previous breast or ovarian cancer, but must be at least one year out from treatment of a Stage 1 or early 2 cancer.

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with high risk of breast cancer
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2001-11; Primary Completion 2006-07 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James M Ford, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States